CLINICAL TRIAL: NCT05413369
Title: A Randomized, 24 Weeks, Active-controlled, Open-label, 2-arm Multicenter Study Comparing the Efficacy and Safety of iGlarLixi to IDegAsp in Chinese Type 2 Diabetes Mellitus Participants Insufficiently Controlled With Oral Antidiabetic Drug(s)
Brief Title: iGlarLixi vs IDegAsp in Chinese Participants After OAD(s)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LPS17396; U1111-1267-2772 (Registry Identifier: ICTRP)
Record Dates: First submitted 2022-06-07; First posted 2022-06-10 (Actual); Results first posted 2024-10-30 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine; lixisenatide; Metformin; Sodium-Glucose Transporter 2 Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- iGlarLixi (Experimental): Participants self-administered iGlarLixi (100 units per milliliter [U/mL] insulin glargine + 100 or 50 microgram [mcg]/mL lixisenatide respectively) subcutaneous (SC) injection once daily on top of metformin +/- sodium-glucose co-transporter 2 inhibitor (SGLT-2i) for 24 weeks. Dose was individually adjusted.
  Interventions: Drug: Insulin glargine/Lixisenatide; Drug: Metformin; Drug: SGLT2 inhibitor
- IDegAsp (Active Comparator): Participants self-administered IDegAsp (100 U/mL of insulin degludec + insulin aspart with a ratio of 70:30) SC injection once daily on top of metformin +/- SGLT-2i for 24 weeks. Dose was individually adjusted.
  Interventions: Drug: IDegAsp; Drug: Metformin; Drug: SGLT2 inhibitor

INTERVENTIONS:
Drug: Insulin glargine/Lixisenatide — solution, by subcutaneous injection
  Arms: iGlarLixi
Drug: IDegAsp — solution, by subcutaneous injection
  Arms: IDegAsp
Drug: Metformin — Tablet, orally
Drug: SGLT2 inhibitor — Tablet, orally

SUMMARY:
This was a parallel-group treatment, Phase 3, randomized, 2-arm study that assessed the efficacy and safety of iGlarLixi to IDegAsp in Chinese T2DM participants insufficiently controlled with oral antidiabetic drug(s).

Study details included:

* Study duration per participant: approximately up to 27 weeks
* Treatment duration: 24 weeks
* Visit frequency: after screening (an on-site visit), on-site or phone call visit every 1 week from randomization till Week 4, every 2 weeks till week 12 and then every 3 weeks till Week 24 (End of Treatment). There were 14 visits that included 7 phone calls and 7 on-site visits in total during screening and treatment periods. There was a safety follow-up by a phone call visit (End of Study) in 3 days after the last dose of the treatment.
* Health measurement/Observation: change in HbA1c as the primary endpoint.
* Intervention name: iGlarLixi and IDegAsp
* Participant sex: male and female
* Participant age range: adults at least 18 years of age
* Condition/disease: Type 2 diabetes mellitus

DETAILED DESCRIPTION:
27 weeks

ELIGIBILITY:
Inclusion Criteria:

* Participant had at least 18 of age inclusive, at the time of signing the informed consent.
* Participants who were diagnosed with T2DM for at least 1 year before the screening visit
* Participants who were treated for at least 3 months prior to the screening visit with a stable dose of metformin (at least 1000 mg/day or the maximum tolerated dose) alone or in combination with a second oral antidiabetic treatment that can be a sulfonylurea (SU), a glinide, an alpha-glucosidase inhibitor (alpha-GI), a dipeptidyl-peptidase-4 (DPP-4) inhibitor or a sodium-glucose co-transporter 2 (SGLT-2) inhibitor
* HbA1c at screening visit:

  * between 7.5% and 11%, both inclusive, for participants previously treated with metformin alone or + SGLT-2 inhibitor, or
  * between 7.0% and 10%, both inclusive, for participants previously treated with metformin + a second oral antidiabetic treatment other than SGLT-2 inhibitor.
* Participants who were overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring.
* Body mass index (BMI) <40 kg/m² at screening
* Male or female, including females of childbearing potential who agreed to use contraception during the study duration
* Participants were capable of giving signed informed consent as described in Appendix 1 of the protocol which included compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

* Participant who had a severe renal function impairment with an estimated glomerular filtration rate (eGFR) <30 mL/min/1.73 m²
* Pregnant or breast-feeding woman.
* Woman of childbearing potential not protected by highly effective contraceptive method of birth control and/or who is unwilling or unable to be tested for pregnancy
* Conditions/situations such as:

  * Participant with short life expectancy.
  * Participant with conditions/concomitant diseases making him/her not evaluable for the primary efficacy endpoint (eg, hemoglobinopathy or hemolytic anemia, receipt of blood or plasma products within 3 months prior to screening).
  * Participant with conditions/concomitant diseases precluding his/her safe participation in this study (eg, active malignant tumor, major systemic diseases, presence of clinically significant diabetic retinopathy or presence of macular edema likely to require laser treatment within the study period).
  * Uncooperative or any condition that could make the participant potentially non-compliant to the study procedures (e.g., participant unable or unwilling to do self-injections or blood glucose monitoring using the Sponsor-provided blood glucometer at home).
* Previous treatment with insulin (except for short-term treatment ≤14 days due to intercurrent illness at the discretion of the Investigator) within 1 year prior to screening.
* Use of oral or injectable glucose-lowering agents other than those stated in the inclusion criteria within 3 months prior to screening.
* Use of systemic glucocorticoids (excluding topical application or inhaled forms) for 1 week or more within 3 months prior to screening.
* Use of weight loss drugs within 3 months prior to screening.
* History of discontinuation of a previous treatment with GLP-1 RAs due to safety/tolerability reasons or lack of efficacy.
* Use of any investigational drug other than specified in this protocol within 1 month or 5 half-lives, whichever is longer, prior to screening.
* Laboratory findings tested at the screening visit:

  * Amylase and/or lipase >3 times the upper limit of normal (ULN) laboratory range.
  * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >3 ULN.
  * Total bilirubin >1.5 ULN (except in case of Gilbert's syndrome).
  * Calcitonin ≥20 pg/mL (5.9 pmol/L).
  * Hemoglobin <10.5 g/dL and/or neutrophils <1500/mm^3 and/or platelets <100 000/mm^3.
  * Positive urine pregnancy test in female of childbearing potential.
* Contraindication to metformin and/or SGLT-2 inhibitor use, for those who were taking it prior to the study, according to local labeling, warning/precaution of use (when appropriate) as displayed in the respective National regulation
* Individuals accommodated in an institution because of regulatory or legal order; prisoners or participants who are legally institutionalized
* Participant not suitable for participation, whatever the reason, as judged by the Investigator, including medical or clinical conditions, or participants potentially at risk of noncompliance to study procedures
* Participants are employees of the clinical study site or other individuals directly involved in the conduct of the study, or immediate family members of such individuals (in conjunction with section 1.61 of the ICH-GCP Ordinance E6)
* Any specific situation during study implementation/course that may raise ethics considerations
* Sensitivity to any of the study interventions (insulin or, or components thereof, or drug or other allergy that, in the opinion of the Investigator, contraindicates participation in the study
* Participants who withdrawn consent at randomization or were lost to follow up at randomization visit.

The above information was not intended to contain all considerations relevant to a potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 582 (Actual)
Dates: Start 2022-07-07 (Actual); Primary Completion 2023-10-20 (Actual); Study Completion 2023-10-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (60):
- China (60):
  - Investigational Site Number : 1560008, Baotou
  - Investigational Site Number : 1560001, Beijing
  - Investigational Site Number : 1560027, Beijing
  - Investigational Site Number : 1560019, Beijing
  - Investigational Site Number : 1560023, Cangzhou
  - Investigational Site Number : 1560059, Changchun
  - Investigational Site Number : 1560046, Changchun
  - Investigational Site Number : 1560052, Changde
  - Investigational Site Number : 1560011, Changsha
  - Investigational Site Number : 1560054, Chengdu
  - Investigational Site Number : 1560024, Chengdu
  - Investigational Site Number : 1560004, Chenzhou
  - Investigational Site Number : 1560044, Chongqing
  - Investigational Site Number : 1560053, Dalian
  - Investigational Site Number : 1560030, Foshan
  - Investigational Site Number : 1560043, Guangzhou
  - Investigational Site Number : 1560029, Guangzhou
  - Investigational Site Number : 1560021, Handan
  - Investigational Site Number : 1560010, Hangzhou
  - Investigational Site Number : 1560045, Harbin
  - Investigational Site Number : 1560025, Harbin
  - Investigational Site Number : 1560038, Hohhot
  - Investigational Site Number : 1560056, Huai'an
  - Investigational Site Number : 1560035, Huanggang
  - Investigational Site Number : 1560055, Huangshi
  - Investigational Site Number : 1560022, Huizhou
  - Investigational Site Number : 1560051, Huzhou
  - Investigational Site Number : 1560040, Jinan
  - Investigational Site Number : 1560014, Jinan
  - Investigational Site Number : 1560058, Jingzhou
  - Investigational Site Number : 1560041, Kaifeng
  - Investigational Site Number : 1560039, Lanzhou
  - Investigational Site Number : 1560060, Lianyungang
  - Investigational Site Number : 1560031, Luoyang
  - Investigational Site Number : 1560028, Nanjing
  - Investigational Site Number : 1560017, Nanjing
  - Investigational Site Number : 1560018, Nanjing
  - Investigational Site Number : 1560057, Nantong
  - Investigational Site Number : 1560037, Pingxiang
  - Investigational Site Number : 1560048, Qingdao
  - Investigational Site Number : 1560012, Qinhuangdao
  - Investigational Site Number : 1560003, Shanghai
  - Investigational Site Number : 1560020, Shanghai
  - Investigational Site Number : 1560007, Shanghai
  - Investigational Site Number : 1560006, Shanghai
  - Investigational Site Number : 1560009, Shenyang
  - Investigational Site Number : 1560050, Suzhou
  - Investigational Site Number : 1560016, Tianjin
  - Investigational Site Number : 1560013, Tianjin
  - Investigational Site Number : 1560047, Tonghua
  - Investigational Site Number : 1560042, Xingtai
  - Investigational Site Number : 1560015, Xuzhou
  - Investigational Site Number : 1560033, Yueyang
  - Investigational Site Number : 1560032, Yueyang
  - Investigational Site Number : 1560026, Yuncheng
  - Investigational Site Number : 1560049, Zhengzhou
  - Investigational Site Number : 1560034, Zhenjiang
  - Investigational Site Number : 1560036, Zhongshan
  - Investigational Site Number : 1560005, Zhuzhou
  - Investigational Site Number : 1560002, Zigong

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: LPS17396 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=25298&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 60 centers in China. A total of 733 participants were screened between 07-Jul-2022 and 17-Apr-2023, of which 151 were screen failures. Screen failures were mainly due to not meeting eligibility criteria.
Pre-assignment Details: A total of 582 participants were randomized in a 1:1 ratio to receive either insulin glargine/lixisenatide (iGlarLixi) or insulin degludec and insulin aspart (IDegAsp).
Period: Overall Study
Arm/Group | iGlarLixi | IDegAsp
Started (Randomized) | 291 | 291
Randomized and Treated | 290 | 291
Completed 24-week Treatment Period | 272 | 284
Completed (Completed the study per protocol) | 274 | 284
Not Completed | 17 | 7
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 13 | 4
Not completed — Non-compliance with study schedule | 2 | 1
Not completed — Other | 1 | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were assessed for all randomized population.
Groups:
- iGlarLixi: Participants self-administered iGlarLixi (100 U/mL insulin glargine + 100 or 50 mcg/mL lixisenatide respectively) SC injection once daily on top of metformin +/- SGLT-2i for 24 weeks. Dose was individually adjusted.
- Total: Total of all reporting groups
Arm/Group | iGlarLixi | IDegAsp | Total
Number analyzed (Participants) | 291 | 291 | 582
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.3 (10.2) | 57.5 (9.9) | 56.9 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 141 | 136 | 277
  Male | 150 | 155 | 305
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 291 | 291 | 582
Glycated Hemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of HbA1c] | 8.58 (0.93) | 8.53 (0.90) | 8.55 (0.91)
Duration of type 2 diabetes [Mean (Standard Deviation); unit: years] | 8.56 (5.68) | 9.06 (6.00) | 8.81 (5.84)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms/square meter (kg/m^2)] | 25.92 (3.47) | 25.42 (3.25) | 25.67 (3.37)
Randomization stratum of oral antidiabetic (OAD) (s) use at screening [Count of Participants; unit: Participants]
  Metformin ± SGLT-2i | 151 | 151 | 302
  Metformin + other OAD | 140 | 140 | 280
  Prior use of SGLT-2i | 37 | 37 | 74

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c From Baseline to Week 24: Non-Inferiority Analysis
Description: Blood samples were collected at indicated timepoints for analysis of HbA1c. Baseline was defined as the last available pre-dose assessment (on or before Day 1).
Time Frame: Baseline, Week 24
Population: Analysis was performed on all randomized participants.
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | iGlarLixi | IDegAsp
Number analyzed (Participants) | 291 | 291
percentage of HbA1c | -1.88 (0.05) | -1.68 (0.05)
Statistical Analysis 1: Comparison: iGlarLixi vs IDegAsp; Statistical analysis for change from baseline in HbA1c; Test type: Non-Inferiority — The non-inferiority was assessed using the upper bound of the 2-sided 95% confidence interval (CI). Non-inferiority p-value was calculated from a non-inferiority margin of 0.3%; p < 0.001, ANCOVA; Treatment groups and randomization stratum of previous oral anti-diabetic drug(OADs) as fixed effects,and baseline HbA1c continuous value as covariate; Least Squares (LS) Mean Difference = -0.20, 95% CI 2-sided [-0.33 to -0.07], Standard Error of Mean 0.07

2. Secondary Outcome: Change in HbA1c From Baseline to Week 24: Superiority Analysis
Description: as for outcome 1
Time Frame: Baseline, Week 24
Population: Analysis was performed on all randomized participants.
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | iGlarLixi | IDegAsp
Number analyzed (Participants) | 291 | 291
percentage of HbA1c | -1.88 (0.05) | -1.68 (0.05)
Statistical Analysis 1: Comparison: iGlarLixi vs IDegAsp; Statistical analysis for change from baseline in HbA1c; Test type: Superiority; p = 0.003, ANCOVA; Treatment groups and randomization stratum of previous as fixed effects, and baseline HbA1c continuous value as covariate; LS Mean Difference = -0.20, 97.5% CI 2-sided [-0.35 to -0.05], Standard Error of Mean 0.07

3. Secondary Outcome: Change in Body Weight From Baseline to Week 24
Description: Body weight was obtained with the participant wearing undergarments or very light clothing and no shoes, and with an empty bladder. The same scale was used throughout the study. Baseline was defined as the last available pre-dose assessment (on or before Day 1).
Time Frame: Baseline, Week 24
Population: Analysis was performed on all randomized participants.
Measure: Least Squares Mean (Standard Error); unit: kilogram
Arm/Group | iGlarLixi | IDegAsp
Number analyzed (Participants) | 291 | 291
kilogram | -0.30 (0.29) | 1.19 (0.25)
Statistical Analysis 1: Comparison: iGlarLixi vs IDegAsp; Statistical analysis for change from baseline in body weight; Test type: Superiority; p < 0.001, ANCOVA; Treatment groups, randomization stratums of HbA1c and previous OADs as fixed effects, and baseline body weight continuous value as covariate; LS Mean Difference = -1.49, 97.5% CI 2-sided [-2.32 to -0.66], Standard Error of Mean 0.37

4. Secondary Outcome: Percentage of Participants Reaching HbA1c <7% at Week 24
Description: Blood samples were collected at indicated timepoints for analysis of HbA1c. Participants without Week 24 HbA1c value were considered as non-responders. Percentages are rounded off to the tenth decimal place.
Time Frame: Week 24
Population: Analysis was performed on all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | iGlarLixi | IDegAsp
Number analyzed (Participants) | 291 | 291
percentage of participants | 72.5 | 59.8
Statistical Analysis 1: Comparison: iGlarLixi vs IDegAsp; Statistical analysis for percentage of participants reaching HbA1c value <7% at Week 24; Test type: Superiority; p < 0.001, Regression, Logistic; Adjusted for treatment group, randomization stratum of previous OADs, and continuous baseline value of HbA1c; Odds Ratio (OR) = 1.89, 97.5% CI 2-sided [1.25 to 2.85]

5. Secondary Outcome: Percentage of Participants Reaching HbA1c <7% With no Body Weight Gain at Week 24
Description: Blood samples were collected at indicated timepoints for analysis of HbA1c. Participants without Week 24 HbA1c or body weight value were considered as non-responders. Percentages are rounded off to the tenth decimal place.
Time Frame: Week 24
Population: Analysis was performed on all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | iGlarLixi | IDegAsp
Number analyzed (Participants) | 291 | 291
percentage of participants | 40.5 | 21.3
Statistical Analysis 1: Comparison: iGlarLixi vs IDegAsp; Statistical analysis for percentage of participants reaching HbA1c value <7% with no body weight gain at Week 24; Test type: Superiority; p < 0.001, Regression, Logistic; Adjusted for treatment group, randomization stratum of previous OADs, and continuous baseline value of HbA1c and body weight; Odds Ratio (OR) = 2.59, 95% CI 2-sided [1.79 to 3.76]

6. Secondary Outcome: Percentage of Participants Reaching HbA1c <7% With no Body Weight Gain at Week 24 and no Hypoglycemia During 24-Week Treatment Period
Description: Blood samples were collected at indicated timepoints for analysis of HbA1c. Participants without Week 24 HbA1c or body weight value were considered as non-responders. During the study, participants were instructed to document the presence of hypoglycemic episodes in their study diary. Hypoglycemia was characterized as per American Diabetes Association (ADA) 2021 recommendations.
  * ADA Level 1 hypoglycemia: A measurable glucose concentration <70 milligram/deciliter (mg/dL) (3.9 millimoles/liter [mmol/L]) but >=54 mg/dL (3.0 mmol/L).
  * ADA Level 2 hypoglycemia: Blood glucose concentration <54 mg/dL [3.0 mmol/L]; the threshold at which neuroglycopenic symptoms begin to occur and requires immediate action to resolve the hypoglycemic event.
  * ADA Level 3 hypoglycemia: A severe event characterized by altered mental and/or physical functioning that requires assistance from another person for recovery.
  Percentages are rounded off to the tenth decimal place.
Time Frame: Baseline up to Week 24
Population: Analysis was performed on all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | iGlarLixi | IDegAsp
Number analyzed (Participants) | 291 | 291
percentage of participants | 26.5 | 13.4
Statistical Analysis 1: Comparison: iGlarLixi vs IDegAsp; Statistical analysis for percentage of participants reaching HbA1c value <7% with no body weight gain at Week 24 and no hypoglycemia during treatment; Test type: Superiority; p < 0.001, Regression, Logistic; [statistical method as in outcome 5, analysis 1]; Odds Ratio (OR) = 2.34, 95% CI 2-sided [1.52 to 3.60]

7. Secondary Outcome: Change in Fasting Plasma Glucose From Baseline to Week 24
Description: Blood samples were collected at fasting state (no food or drinks [except water] for at least 8 hours) at indicated timepoints. Baseline was defined as the last available pre-dose assessment (on or before Day 1).
Time Frame: Baseline, Week 24
Population: Analysis was performed on all randomized participants.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | iGlarLixi | IDegAsp
Number analyzed (Participants) | 291 | 291
mmol/L | -3.18 (0.11) | -3.45 (0.11)

8. Secondary Outcome: Change in Average 7-Point Self-Monitored Plasma Glucose (SMPG) Profile From Baseline to Week 24
Description: Participants were provided with a glucometer, corresponding supplies, a leaflet, and with diaries in order to perform self-measurement of plasma glucose and its recording and were trained on how to use the glucometer. The 7-point SMPG profile was measured at the following 7-points: pre-prandial (before starting a meal) and 2 hours postprandial each for breakfast, lunch, dinner and at bedtime. Two hours postprandial (breakfast, lunch and dinner) was defined as 2 hours after the start of the meal. The participants performed 7-point SMPG profile measurement over a single 24-hour period on 2 different days in the week. Baseline was defined as the last available pre-dose assessment (on or before Day 1).
Time Frame: Baseline, Week 24
Population: Analysis was performed on all randomized participants.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | iGlarLixi | IDegAsp
Number analyzed (Participants) | 291 | 291
mmol/L | -3.36 (0.12) | -2.92 (0.11)

9. Secondary Outcome: Percentage of Participants Reaching HbA1c <7% at Week 24 With no Hypoglycemia During 24-Week Treatment Period
Description: Blood samples were collected at indicated timepoints for analysis of HbA1c. Participants without Week 24 HbA1c value were considered as non-responders. Hypoglycemia was characterized as per ADA 2021 recommendations.
  * ADA Level 1 hypoglycemia: A measurable glucose concentration <70 mg/dL (3.9 mmol/L) but >=54 mg/dL (3.0 mmol/L).
  * ADA Level 2 hypoglycemia: Blood glucose concentration <54mg/dL [3.0 mmol/L]; the threshold at which neuroglycopenic symptoms begin to occur and requires immediate action to resolve the hypoglycemic event.
  * ADA Level 3 hypoglycemia: A severe event characterized by altered mental and/or physical functioning that requires assistance from another person for recovery.
  Percentages are rounded off to the tenth decimal place.
Time Frame: Baseline up to Week 24
Population: Analysis was performed on all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | iGlarLixi | IDegAsp
Number analyzed (Participants) | 291 | 291
percentage of participants | 43.6 | 35.7

10. Secondary Outcome: Percentage of Participants Reaching HbA1c <7% at Week 24 With no Clinically Relevant Hypoglycemia During 24-Week Treatment Period
Description: Blood samples were collected at indicated timepoints for analysis of HbA1c. Participants without Week 24 HbA1c value were considered as non-responders. Participants who reached the specified target of HbA1c without any clinically significant symptoms of hypoglycemia as defined in ADA Levels 2 or 3 are reported. Percentages are rounded off to the tenth decimal place.
Time Frame: Baseline up to Week 24
Population: Analysis was performed on all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | iGlarLixi | IDegAsp
Number analyzed (Participants) | 291 | 291
percentage of participants | 66.7 | 56.0

11. Secondary Outcome: Total Daily Insulin Dose at Week 24
Description: Total daily insulin dose was defined as the sum of the insulin dose from study treatment and non-study treatment (e.g., rescue therapy). It was the average of the last 3 available insulin doses recorded in the electronic case report form in the week before visit.
Time Frame: Week 24
Population: Analysis was performed on all randomized participants.
Measure: Least Squares Mean (Standard Error); unit: units
Arm/Group | iGlarLixi | IDegAsp
Number analyzed (Participants) | 291 | 291
units | 27.68 (0.84) | 33.78 (0.83)

12. Secondary Outcome: Percentage of Participants Who Required Rescue Therapy During the 24-Week Treatment Period
Description: Routine HbA1c value was used to determine the requirement of rescue medication. Threshold value was HbA1c >8% at Week 12 or later on despite appropriate corrective actions. Percentages are rounded off to the tenth decimal place.
Time Frame: Baseline up to Week 24
Population: Analysis was performed on all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | iGlarLixi | IDegAsp
Number analyzed (Participants) | 291 | 291
percentage of participants | 5.2 | 6.9

13. Secondary Outcome: Change in Fasting C-Peptide From Baseline to Week 24
Description: as for outcome 7
Time Frame: Baseline, Week 24
Population: Analysis was performed on all randomized participants. Only those participants with data collected at baseline and Week 24 are reported.
Measure: Least Squares Mean (Standard Error); unit: nanomoles/liter (nmol/L)
Arm/Group | iGlarLixi | IDegAsp
Number analyzed (Participants) | 190 | 196
nanomoles/liter (nmol/L) | -0.23 (0.02) | -0.33 (0.02)

14. Secondary Outcome: Number of Participants With Any Hypoglycemia Event During On-Treatment Period
Description: During the study, participants were instructed to document the presence of hypoglycemic episodes in their study diary. Number of participants who met ADA definition of hypoglycemia during the treatment period are reported.
  * ADA Level 1 hypoglycemia: A measurable glucose concentration <70 mg/dL (3.9 mmol/L) but >=54 mg/dL (3.0 mmol/L).
  * ADA Level 2 hypoglycemia: Blood glucose concentration <54mg/dL [3.0 mmol/L]; the threshold at which neuroglycopenic symptoms begin to occur and requires immediate action to resolve the hypoglycemic event.
  * ADA Level 3 hypoglycemia: A severe event characterized by altered mental and/or physical functioning that requires assistance from another person for recovery.
  The on-treatment period (ie, treatment-emergent [TE] period) was defined as the period from the first injection study treatment to the last injection of study treatment + 3 days (1 day for hypoglycemia).
Time Frame: From first dose of study drug up to 1 day after the last administration of study drug (maximum treatment exposure: 192 days)
Population: Analysis was performed on safety population which included all randomized participants who had taken at least 1 dose of study intervention, regardless of the amount of treatment administered.
Measure: Count of Participants; unit: Participants
Arm/Group | iGlarLixi | IDegAsp
Number analyzed (Participants) | 290 | 291
Participants | 102 | 118

15. Secondary Outcome: Hypoglycemic Event Rate During the On-Treatment Period
Description: During the study, participants were instructed to document the presence of hypoglycemic episodes in their study diary. Percentage of hypoglycemic events per participant-year during on-treatment period are reported. The on-treatment period (TE period) was defined as the period from the first injection study treatment to the last injection of study treatment + 3 days (1 day for hypoglycemia).
Time Frame: as for outcome 14
Population: Analysis was performed on safety population.
Measure: Number; unit: event rate per participant-year
Arm/Group | iGlarLixi | IDegAsp
Number analyzed (Participants) | 290 | 291
event rate per participant-year | 1.90 | 2.72

16. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Treatment-Emergent Serious Adverse Events (TESAEs), Adverse Events Of Special Interest (AESIs) and TEAEs Leading to Treatment Discontinuation
Description: An AE was any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An SAE was defined as any adverse event that, at any dose resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect or was a suspected transmission of any infectious agent via an authorized medicinal product. An AESI was an AE (serious or nonserious) of scientific and medical concern specific to the Sponsor's product or program, for which ongoing monitoring and immediate notification by the Investigator to the Sponsor was required. TE period was defined as the period from the first injection study treatment to the last injection of study treatment + 3 days.
Time Frame: From signature of the informed consent form up to the final visit regardless of seriousness or relationship to study drug (maximum treatment exposure: 192 days)
Population: Analysis was performed on the safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | iGlarLixi | IDegAsp
Number analyzed (Participants) | 290 | 291
Participants
  Any TEAE | 220 | 192
  Any TESAE | 15 | 12
  Any AESI | 6 | 2
  Any TEAE leading to treatment discontinuation | 7 | 1

17. Secondary Outcome: Number of Participants With Potentially Clinically Significant Laboratory Abnormalities (PCSA): Vital Signs
Description: Vital signs assessments included systolic blood pressure (SBP), diastolic blood pressure (DBP) and heart rate (HR) in sitting position with their arm outstretched in line with mid-sternum and supported and weight. Criteria for PCSA: SBP: <=95 millimeters of mercury (mmHg) and decrease from baseline >=20 mmHg, >=160 mmHg and increase from baseline >=20 mmHg; DBP :<=45 mmHg and decrease from baseline >=10 mmHg,>=110 mmHg and increase from baseline >=10 mmHg; HR: <=50 beats/min and decrease from baseline >=20 beats/min,>=120 beats/min and increase from baseline >=20 beats/min; Weight >=5% decrease from baseline, >=5% increase from baseline.
Time Frame: From first dose of study drug up to 3 days after last administration of study drug (maximum treatment exposure: 192 days)
Population: Analysis was performed on the safety population. Only those participants with data collected for each parameter during TE period are reported.
Measure: Count of Participants; unit: Participants
Arm/Group | iGlarLixi | IDegAsp
Number analyzed (Participants) | 290 | 291
Participants
  SBP: <=95 mmHg and decrease from baseline >=20 mmHg: number analyzed (Participants) | 288 | 290
  SBP: <=95 mmHg and decrease from baseline >=20 mmHg | 1 | 1
  SBP: >=160 mmHg and increase from baseline >=20 mmHg: number analyzed (Participants) | 288 | 290
  SBP: >=160 mmHg and increase from baseline >=20 mmHg | 4 | 7
  DBP :<=45 mmHg and decrease from baseline >=10 mmHg: number analyzed (Participants) | 288 | 290
  DBP :<=45 mmHg and decrease from baseline >=10 mmHg | 0 | 0
  DBP: >=110 mmHg and increase from baseline >=10 mmHg: number analyzed (Participants) | 288 | 290
  DBP: >=110 mmHg and increase from baseline >=10 mmHg | 0 | 0
  HR: <=50 beats/min and decrease from baseline >=20 beats/min: number analyzed (Participants) | 288 | 290
  HR: <=50 beats/min and decrease from baseline >=20 beats/min | 0 | 0
  HR: >=120 beats/min and increase from baseline >=20 beats/min: number analyzed (Participants) | 288 | 290
  HR: >=120 beats/min and increase from baseline >=20 beats/min | 0 | 0
  Weight: >=5% decrease from baseline: number analyzed (Participants) | 288 | 290
  Weight: >=5% decrease from baseline | 41 | 19
  Weight: >=5% increase from baseline: number analyzed (Participants) | 288 | 290
  Weight: >=5% increase from baseline | 29 | 73

18. Secondary Outcome: Number of Participants With Potentially Clinically Significant Laboratory Abnormalities (PCSA): Hematology
Description: Criteria for PCSA: For Hemoglobin (Hb), there are 3 criteria: (1)<=115 grams (g)/L (Male[M]) or <=95 g/L (Female[F]), (2)>= 185 g/L (M) or >=165 g/L (F), and (3) decrease from baseline >=20 g/L; Hematocrit: <=0.37 volume/volume (v/v) (M) or <=0.32 v/v (F), >=0.55 v/v (M) or >=0.5 v/v (F); Red blood cells (RBC): >=6 Tera/L; Platelets: <100 Giga/L, >=700 Giga/L; White blood cells (WBC): <3.0 Giga/L (Non-Black [NB]); <2.0 Giga/L (Black [B]) or >=16.0 Giga/L; Neutrophils: <1.5 Giga/L (NB) or <1.0 Giga/L (B); Lymphocytes: >4.0 Giga/L; Monocytes: >0.7 Giga/L; Basophils: >0.1 Giga/L; Eosinophils: >0.5 Giga/L or >upper limit of normal (ULN) (if ULN >=0.5 Giga/L).
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | iGlarLixi | IDegAsp
Number analyzed (Participants) | 290 | 291
Participants
  Hb: <=115 g/L (M); <=95 g/L (F): number analyzed (Participants) | 285 | 288
  Hb: <=115 g/L (M); <=95 g/L (F) | 4 | 1
  Hb: >=185 g/L (M); >=165 g/L (F): number analyzed (Participants) | 285 | 288
  Hb: >=185 g/L (M); >=165 g/L (F) | 1 | 4
  Hb: Decrease from Baseline >=20 g/L: number analyzed (Participants) | 285 | 288
  Hb: Decrease from Baseline >=20 g/L | 25 | 19
  Hematocrit: <=0.37 v/v (M) or <=0.32 v/v (F): number analyzed (Participants) | 285 | 288
  Hematocrit: <=0.37 v/v (M) or <=0.32 v/v (F) | 2 | 6
  Hematocrit: >=0.55 v/v (M) or >=0.5 v/v (F): number analyzed (Participants) | 285 | 288
  Hematocrit: >=0.55 v/v (M) or >=0.5 v/v (F) | 37 | 30
  RBC: >=6 Tera/L: number analyzed (Participants) | 285 | 288
  RBC: >=6 Tera/L | 5 | 6
  Platelets: <100 Giga/L: number analyzed (Participants) | 284 | 288
  Platelets: <100 Giga/L | 3 | 7
  Platelets: >=700 Giga/L | 0 | 0
  WBC: <3.0 Giga/L (NB); < 2.0 Giga/L (B): number analyzed (Participants) | 285 | 288
  WBC: <3.0 Giga/L (NB); < 2.0 Giga/L (B) | 2 | 3
  WBC: >=16.0 Giga/L: number analyzed (Participants) | 285 | 288
  WBC: >=16.0 Giga/L | 1 | 0
  Neutrophils: <1.5 Giga/L (NB) or <1.0 Giga/L (B): number analyzed (Participants) | 285 | 288
  Neutrophils: <1.5 Giga/L (NB) or <1.0 Giga/L (B) | 5 | 7
  Lymphocytes: > 4.0 Giga/L: number analyzed (Participants) | 285 | 288
  Lymphocytes: > 4.0 Giga/L | 4 | 6
  Monocytes: >0.7 Giga/L: number analyzed (Participants) | 285 | 288
  Monocytes: >0.7 Giga/L | 35 | 29
  Basophils: >0.1 Giga/L: number analyzed (Participants) | 285 | 288
  Basophils: >0.1 Giga/L | 2 | 5
  Eosinophils: >0.5 Giga/L or >ULN: number analyzed (Participants) | 285 | 288
  Eosinophils: >0.5 Giga/L or >ULN | 2 | 2

19. Secondary Outcome: Number of Participants With Potentially Clinically Significant Laboratory Abnormalities (PCSA): Clinical Chemistry
Description: Criteria for PCSA: Lipase: >=3 ULN; Amylase: >=3 ULN; Sodium: <=129 mmol/L; >=160 mmol/L; Potassium: <3 mmol/L, >=5.5 mmol/L; Creatinine: >=150 micromoles per liter (umol/L), >=30% or >=100% change from baseline; Glomerular filtration rate (GFR): >=60-<90 mL/minute(min)/1.73 square meter (m^2) (mild decrease in GFR), >=30-<60 mL/min/1.73m^2 (moderate decrease in GFR), >=15-<30 mL/min/1.73m^2 (severe decrease in GFR),<15 mL/min/1.73m^2 (end stage renal disease); Creatinine clearance (CG): >=60-<90 mL/min (mild decrease in GFR), >=30-<60 mL/min (moderate decrease in GFR), >=15-<30 mL/min (severe decrease in GFR), <15 mL/min (end stage renal disease); Urea nitrogen (BUN): >=17 mmol/L and Uric acid: <120 or >408 umol/L; Alanine transaminase (ALT) and aspartate transaminase (AST): >3/5/10/20 ULN. Alkaline phosphatase:>1.5 ULN, total bilirubin (TBILI): >1.5 or >2 ULN, ALT and TBILI:> ALT>3ULN and TBILI >2 ULN and Conjugated and total bilirubin: >35% TBILI and TBILI >1.5 ULN.
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | iGlarLixi | IDegAsp
Number analyzed (Participants) | 290 | 291
Participants
  Lipase: >=3 ULN: number analyzed (Participants) | 285 | 288
  Lipase: >=3 ULN | 6 | 9
  Amylase: >=3 ULN | 0 | 0
  Sodium: <=129 mmol/L | 0 | 0
  Sodium: >=160 mmol/L | 0 | 0
  Potassium: <3 mmol/L | 0 | 0
  Potassium: >=5.5 mmol/L: number analyzed (Participants) | 285 | 288
  Potassium: >=5.5 mmol/L | 1 | 3
  Creatinine: >=150 umol/L: number analyzed (Participants) | 285 | 288
  Creatinine: >=150 umol/L | 0 | 1
  Creatinine: >=30% change from baseline: number analyzed (Participants) | 285 | 288
  Creatinine: >=30% change from baseline | 36 | 29
  Creatinine: >=100% change from baseline: number analyzed (Participants) | 285 | 288
  Creatinine: >=100% change from baseline | 0 | 1
  GFR: Mild decrease in GFR: number analyzed (Participants) | 285 | 288
  GFR: Mild decrease in GFR | 80 | 79
  GFR: Moderate decrease in GFR: number analyzed (Participants) | 285 | 288
  GFR: Moderate decrease in GFR | 11 | 11
  GFR: Severe decrease in GFR: number analyzed (Participants) | 285 | 288
  GFR: Severe decrease in GFR | 0 | 1
  GFR: End stage renal disease | 0 | 0
  CG: Mild decrease in GFR: number analyzed (Participants) | 285 | 288
  CG: Mild decrease in GFR | 80 | 85
  CG: Moderate decrease in GFR: number analyzed (Participants) | 285 | 288
  CG: Moderate decrease in GFR | 12 | 16
  CG: Severe decrease in GFR | 0 | 0
  CG: End stage renal disease | 0 | 0
  BUN: >=17 mmol/L | 0 | 0
  Uric Acid: <120 umol/L | 0 | 0
  Uric Acid: >408 umol/L: number analyzed (Participants) | 285 | 288
  Uric Acid: >408 umol/L | 104 | 108
  ALT: >3 ULN: number analyzed (Participants) | 285 | 288
  ALT: >3 ULN | 4 | 2
  ALT: >5 ULN: number analyzed (Participants) | 285 | 288
  ALT: >5 ULN | 1 | 0
  ALT: >10 ULN: number analyzed (Participants) | 285 | 288
  ALT: >10 ULN | 1 | 0
  ALT: >20 ULN | 0 | 0
  AST: >3 ULN | 0 | 0
  AST: >5 ULN: number analyzed (Participants) | 285 | 288
  AST: >5 ULN | 1 | 0
  AST: >10 ULN | 0 | 0
  AST: >20 ULN | 0 | 0
  Alkaline Phosphatase: >1.5 ULN: number analyzed (Participants) | 285 | 288
  Alkaline Phosphatase: >1.5 ULN | 2 | 5
  TBILI: >1.5 ULN: number analyzed (Participants) | 285 | 288
  TBILI: >1.5 ULN | 3 | 1
  TBILI: >2 ULN: number analyzed (Participants) | 285 | 288
  TBILI: >2 ULN | 1 | 0
  ALT>3ULN and TBILI >2 ULN | 0 | 0
  Conjugated and TBILI: >35% TBILI and TBILI >1.5 ULN: number analyzed (Participants) | 285 | 288
  Conjugated and TBILI: >35% TBILI and TBILI >1.5 ULN | 2 | 0

ADVERSE EVENTS:
Time Frame: From signature of the informed consent form up to the final visit regardless of seriousness or relationship to study drug (maximum treatment exposure: 192 days). All-cause mortality was collected throughout the study, up to 67 weeks.
Description: Analysis was performed on the safety population.
Arm/Group | iGlarLixi | IDegAsp
All-Cause Mortality (participants affected / at risk) | 0/290 | 0/291
Serious Adverse Events (participants affected / at risk) | 15/290 | 12/291
Other Adverse Events (participants affected / at risk) | 152/290 | 101/291
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | iGlarLixi (N=290) | IDegAsp (N=291)
Bronchopulmonary Aspergillosis (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal Infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Intraosseous Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebral Infarction (Nervous system disorders) | 2 (2) | 1 (1)
Ischaemic Cerebral Infarction (Nervous system disorders) | 1 (1) | 0 (0)
Vertebrobasilar Insufficiency (Nervous system disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Sudden Hearing Loss (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Arteriosclerosis Coronary Artery (Cardiac disorders) | 0 (0) | 1 (1)
Coronary Artery Disease (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial Ischaemia (Cardiac disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Varicophlebitis (Vascular disorders) | 0 (0) | 1 (1)
Lung Disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Gastric Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cholecystitis Acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 1 (1)
Uterine Polyp (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Chest Discomfort (General disorders) | 0 (0) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 1 (1) | 0 (0)
Femur Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Humerus Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | iGlarLixi (N=290) | IDegAsp (N=291)
Covid-19 (Infections and infestations) | 39 (39) | 31 (31)
Upper Respiratory Tract Infection (Infections and infestations) | 50 (60) | 37 (42)
Hyperuricaemia (Metabolism and nutrition disorders) | 26 (31) | 24 (27)
Dizziness (Nervous system disorders) | 19 (21) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 16 (18) | 7 (8)
Nausea (Gastrointestinal disorders) | 35 (50) | 2 (3)
Vomiting (Gastrointestinal disorders) | 15 (17) | 0 (0)
Lipase Increased (Investigations) | 19 (24) | 16 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2022-06-16): https://cdn.clinicaltrials.gov/large-docs/69/NCT05413369/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-14): https://cdn.clinicaltrials.gov/large-docs/69/NCT05413369/SAP_001.pdf